CLINICAL TRIAL: NCT06437912
Title: Effectiveness of Botulinum Toxin A in Preventing Scar Formation and Initial Exploration of "Optimal
Brief Title: Effectiveness of Botulinum Toxin A in Preventing Scar Formation and Initial Exploration of "Optimal Concentration"
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Dezhou Hospital Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MR-37-23-008382
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Scar
Keywords: scar prevention; botulinum toxin type A
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Injection 1 U / 0.1ml BTXA (Experimental): Botulinum toxin type A (BTXA) was injected into both sides of the knife edge immediately after operation, the injection volume was 1U/0.1ml per point, the interval between the injection points on the same side of the knife edge was 1cm, and the distance of each injection point from the knife edge was 0.5cm. It was injected only once immediately after operation.
  Interventions: Drug: Botulinum toxin type A
- Injection 2.5U / 0.1ml BTXA (Experimental): Botulinum toxin type A (BTXA) was injected into both sides of the knife edge immediately after operation, the injection volume was 2.5U/0.1ml per point, the interval between the injection points on the same side of the knife edge was 1cm, and the distance of each injection point from the knife edge was 0.5cm. It was injected only once immediately after operation.
  Interventions: Drug: Botulinum toxin type A
- Injection 5U / 0.1ml BTXA (Experimental): Botulinum toxin type A (BTXA) was injected into both sides of the knife edge immediately after operation, the injection volume was 5U/0.1ml per point, the interval between the injection points on the same side of the knife edge was 1cm, and the distance of each injection point from the knife edge was 0.5cm. It was injected only once immediately after operation.
  Interventions: Drug: Botulinum toxin type A
- Injection 0.9%Nacl (Active Comparator): Injection 0.9%Nacl Immediately after operation 0.9%Nacl was injected on both sides of the knife edge, the injection volume per point was 0.1ml, the interval between each injection point on the same side of the knife edge was 1cm, and each injection point was away from the knife edge 0.5cm. It was injected only once immediately after operation.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Eligible patients were randomly assigned to the experimental group and the control group. Patients in the experimental group will be randomized to receive injections of 1 U,2.5 U, and 5 U botulinum toxin type A,Patients in the control group received an injection of 0.9% Nacl
  Other Names: 0.9%Nacl

SUMMARY:
Each year, millions of burn, trauma, or surgical patients worldwide suffer from scarring that severely affects their quality of life and social functioning. In order to prevent and treat diseases related to abnormal scar hyperplasia, clinicians and researchers have adopted various methods, such as scar grinding, surgical resection, drug injection in scar tissue, cryotherapy, laser and so on. However, these methods can not effectively inhibit the abnormal proliferation of scars and improve the adverse effects of existing scars on patients. To date, there is no accepted gold standard for the effective treatment and improvement of abnormal scar tissue.

DETAILED DESCRIPTION:
Through a large number of literature review and preliminary experiments, we summarized and found the following problems: a. The latest research on prevention of scar formation by botulinum toxin type A is only aimed at surgical wounds from the wound type, and there is no research on the scar prevention effect of trauma wounds. b. From the point of view of the study site, there is no study on the effect of scar prevention only on the head, neck, chest and other parts of the body. c. For the research results of botulinum toxin type A in the prevention of scarring, the current research focuses on the effectiveness of botulinum toxin type A at a certain concentration, and does not compare the effects of botulinum toxin type A at various concentrations.Therefore, in order to explore the "optimal concentration" of botulinum toxin type A to prevent scar formation; To explore the effect of botulinum toxin A on scar prevention of traumatic wounds and surgical incisions. To explore the effect of botulinum toxin A on scar prevention in other parts of the body in addition to effective prevention of head, neck and chest scar, We intend to focus on the effectiveness and "optimal concentration" of botulinum toxin type A to prevent scarring, to determine the effect of this means on scar prevention, to provide new ideas for botul

ELIGIBILITY:
Inclusion Criteria:

Patients with emergency trauma and skin swellings, with clear consciousness, no mental retardation or cognitive difficulties, agree to participate in this study, 12≤ age ≤ 65 years old

Exclusion Criteria:

Allergic to botulinum toxin type A;Pregnant, lactating women, patients who plan to get pregnant in the near future;Patients taking retinoic acid, synthetic steroids, amino glycosides antibiotics, calcium channel blockers, cyclosporine and cholinesterase inhibitors; 4 Neuromuscular diseases: such as myasthenia gravis, Lambert-Eaton syndrome, multiple sclerosis;5. Patients with cardiovascular diseases, kidney diseases, liver and other basic diseases; 6 Patients with infection at the injection site; 7 Expect unrealistic patients.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
The modified Stony Brook Scar Evaluation Scale | Postoperative 7 days, 15 days, 1 month, 3 months, 6 months
  The mSBSES included width (0 = scar enlargement prominent and > 2 mm, 1 = presence of scar enlargement ≤ 2 mm, 2 = no scar widening), height (0 = marked scar uplift, 1 = presence of scar uplift, 2 = no scar uplift), color (0 = scar significantly redder than surrounding, 1 = scar redder than surrounding and 2 = scar the same color as or lighter than surrounding skin), The visibility of the incision line (0 = marked incision line, 1 = presence of incision line, 2 = absence of incision line) was objectively assessed separately in non-chronological order, with overall scar values varying from 0 to 8, with higher scores indicating better scar appearance.

SECONDARY OUTCOMES:
Patient satisfaction and perceptions represented secondary outcome measures in this study | Postoperative 7 days, 15 days, 1 month, 3 months, 6 months
  Patient Satisfaction Scale (1=dissatisfied, 2=slightly satisfied, 3=satisfied, and 4=very satisfied). They were also asked to assess their levels of pain (0=no pain, 1=mild, 2=moderate, 3=severe, 4=very painful) and pruritus (0=no itch, 1=mild, 2=moderate, 3=severe, 4=very itchy) at the incision site. The totals varied between 0-8, where lower scores indicated more positive subjective patient perceptions.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University Dezhou Hospital, Dezhou, Shandong, China

IPD SHARING:
Plan to Share IPD: No